CLINICAL TRIAL: NCT04421313
Title: Supplementation of Rheumatoid Arthritis Patients With Dietary Fibre to Improve Their Gut Microbiota
Brief Title: Fibres Supplementation in Rheumatoid Arthritis
Acronym: SUPER-FIBRES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University of Sydney (Other); Institut de Génétique Moléculaire de Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECHMPL17_0397
Record Dates: First submitted 2020-05-18; First posted 2020-06-09 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; dietary fibre; gut-microbiota; SCFAs
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhumatoid Arthritis (Experimental): The patients with Rheumatoid arthritis receive 12 g/day of INULIN or 10,5g/day of maltodextrine during 30 days
  Interventions: Drug: Dietary Fiber Supplementation
- Control Subjects (Placebo Comparator): The patients with Control Subjects receive 12 g/day of INULIN or 10,5g/day of maltodextrine during 30 days
  Interventions: Drug: Dietary Fiber Supplementation

INTERVENTIONS:
Drug: Dietary Fiber Supplementation — 12 g of inulin or of maltodextrin in powder, to dilute in water once daily, during 1 month. Given in pre-weighted pots (one pot per day, similar color and aspect)

SUMMARY:
Design: Randomized, double-blind, placebo-controlled study with 4 weeks of treatment with either fiber supplements or placebo.

Primary outcome: variation in SCFA between baseline and week 4. Secondary outcomes : variations in gut microbiota, disease activity (DAS28, RAID), immune cells (regulatory T and B cells, Th17) and heart-rate variability.

Population: 29 patients with rheumatoid arthritis treated with only csDMARDs and a moderate disease activity will be recruited in each arm and 29 controls with mechanic disease (osteoarthritis, tendinitis).

Collection: Blood, feces, disease activity and heart rate variability will be collected at baseline and week 4.

ELIGIBILITY:
General

Inclusion criteria:

* Aged 18 to 85
* Be affiliated to or beneficiary of a French social security scheme
* o No desire for pregnancy for the duration of the study (Effective contraception for women of reproductive age, for the duration of the study (surgical sterilization, hormonal contraceptives, barrier method, intrauterine device))

Exclusion criteria:

* Lack of written informed consent after a period of reflection
* Patient involved in other research or research for which the exclusion period has not ended
* Pregnant or nursing woman
* Type I or II diabetes
* Patient receiving more than 10 mg/d corticosteroids at time of inclusion
* Patient who received corticosteroid infusions in the month prior to randomization
* Unusual consumption (>50% higher than usual consumption) of dietary fibre in the last 72 hours (assessed by food questionnaire)

Patient with Rheumatoid polyarthritis

Inclusion criteria:

* Rheumatoid arthritis meeting ACR/EULAR 2010 criteria
* With moderate clinical activity: DAS28-CRP 3.2 and 5.1
* Patient receiving conventional background treatment at stable doses and should not be modified during 4-week follow-up

Exclusion criteria:

* Patient treated by targeted RA treatment in the year prior to inclusion
* Patient who received antibiotic therapy within 3 months prior to randomization

Control subjects

Inclusion criteria:

* Patient consulting in the rheumatology department for a mechanical pathology: osteoarthritis of the limbs or spine, osteoporosis, tendinopathy, fibromyalgia, algodystrophy or capsulitis.
* Matched to a gender and age PR topic 5 years

Exclusion criteria:

· Patient with autoimmune disease, infection or progressive cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Short-chain fatty acid (SCFA) | 36 months

SECONDARY OUTCOMES:
Description of the gut microbiota bacteria | 36 months
  Amplification of the V1-V3 bacterial region targeting 16S bacterial ribosomal RNA and sequencing by Mi-sequencer will be performed. Then, a bioinformatics analysis will be done using the QIIME software and the composition of the intestinal flora will be analyzed.
Description of immune cells (regulatory T and B cells, Th17) | 36 months
  Flow cytometric determination of immune cells
Evaluation of heart-rate variability. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Claire DAIEN, Principal Investigator — CHU of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France